CLINICAL TRIAL: NCT05304962
Title: First-in-Human, Escalating Oral Dose Study of RGT-419B Given Alone and With Endocrine Therapy in Subjects With Hormone Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative Advanced/Metastatic Breast Cancer
Brief Title: FIH Study of RGT-419B Alone and With Endocrine Therapy in HR-Positive, HER2-Negative Advanced/Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regor Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RGT-419B_01-101
Record Dates: First submitted 2022-02-24; First posted 2022-03-31 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: There will be two study arms opened sequentially to the same patient population. Arm A is RGT-419B alone (singlet). Arm B is RGT-419B + Hormonal Therapy (doublet) and will follow completion of Arm A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): RGT-419B given alone as monotherapy
  Interventions: Drug: RGT-419B
- Arm B (Experimental): RGT-419B in combination with Hormonal Therapy
  Interventions: Drug: RGT-419B in combination with hormonal therapy

INTERVENTIONS:
Drug: RGT-419B — oral capsules
  Arms: Arm A
Drug: RGT-419B in combination with hormonal therapy — RGT-419B in combination with hormonal therapy (Selective Estrogen Receptor Degrader, Selective Estrogen Receptor Modulator, or Aromatase Inhibitor)
  Arms: Arm B

SUMMARY:
This is a phase I, First-in-Human (FIH), open-label study to evaluate the safety, tolerability, pharmacokinetic (PK) profile, and preliminary efficacy of RGT-419B administered orally as monotherapy OR in combination with Hormonal Therapy in subjects with HR+, HER2- locally advanced and unresectable (Stage III) or metastatic (Stage IV) breast cancer whose disease has progressed during prior therapy with an approved CDK4/6i plus hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >/= 18 years old
2. ECOG Performance Status 0 to 1
3. Subjects must have histologically or cytologically confirmed diagnosis of ER+, HER2- ABC consistent with ASCO CAP guidelines that is locally advanced and unresectable (Stage III) or metastatic (Stage IV) BC.
4. Measurable AND evaluable lesions at baseline per RECIST v1.1.
5. Eligible subjects must meet all of the following criteria:

   * Progression after receiving 1 line of prior cyclin-dependent kinase 4 and 6 inhibitor (CDK4/6i) therapy combined with HT in the MBC setting (up to 1 additional line of CDK4/6i is permitted in the post-surgical adjuvant setting);

     * Subjects must have received therapy for ≥3 months in the MBC setting, or for ≥6 months in the adjuvant setting, prior to progression
   * Progression after ≤3 lines of prior HT therapy (regardless of whether it is HT alone or in combination with other therapies)

     * Prior HT combination agents, including SERD, SERM or AI, must have received formal approval by regulatory agency.
   * ≤ 1 prior line of chemotherapy in the metastatic setting
6. Adequate organ function
7. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Presence of visceral metastases with severe organ dysfunction as evidence by signs and symptoms, laboratory studies, lymphangitic spread and/or rapid progression of disease
2. Pregnant or planning to become pregnant
3. Prior irradiation to >25% of the bone marrow and/or inadequate bone marrow function or evidence of clinically significant end-organ damage
4. Major surgery, chemotherapy, targeted therapy, experimental agents, or radiation within 14-28 days prior to Cycle 1, Day 1
5. Active, serious medical condition that is not well controlled with locally approved medications allowed by the protocol
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the drugs used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety & Tolerability - Number of subjects with Dose-Limiting Toxicities (DLTs) at each cohort dose level in singlet and doublet therapy | 4 weeks (1 cycle)
  Number of subjects who have a confirmed DLT at each cohort dose level in singlet and doublet study arms during the first 28-day cycle of RGT-419B treatment.

SECONDARY OUTCOMES:
Safety & Tolerability - Incidence, Severity, and Causality of all Treatment Emergent Adverse Events (TEAEs) | through study completion, an average of 1 year
  Incidence, severity, and causality of all TEAEs will be assessed for all patient participating from Day 1 dosing through end of study.
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Cmax | through study completion, an average of 1 year
  Plasma and urine samples that are being collected for PK assessment may also be used for exploratory metabolite identification
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Area Under Concentration-Time Curve (AUC0-t) | through study completion, an average of 1 year
  Plasma and urine samples that are being collected for PK assessment may also be used for exploratory metabolite identification
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Area Under Concentration-Time Curve to Infinity (AUC0-inf) | through study completion, an average of 1 year
  Plasma and urine samples that are being collected for PK assessment may also be used for exploratory metabolite identification
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Plasma Decay Half-Life (t 1/2) | through study completion, an average of 1 year
  Plasma and urine samples that are being collected for PK assessment may also be used for exploratory metabolite identification
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Time to Reach Maximum Observed Plasma Concentration (Tmax) | through study completion, an average of 1 year
  Plasma and urine samples that are being collected for PK assessment may also be used for exploratory metabolite identification
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Accumulation rate after multiple doses | through study completion, an average of 1 year
  Plasma and urine samples that are being collected for PK assessment may also be used for exploratory metabolite identification
Day 1 and steady-state PK assessment of RGT-419B and major metabolites - Cumulative urinary excretion | through study completion, an average of 1 year
  Plasma and urine samples that are being collected for PK assessment may also be used for exploratory metabolite identification
Tumor Response assessed by Investigator according to RECIST v1.1 | through study completion, an average of 1 year
  Tumor response measured by radiologic imaging techniques at baseline and throughout the study
QTc Interval - Changes in corrected QT interval | through study completion, an average of 1 year
  Number of subjects with a clinically significant increase from baseline in corrected QT (QTc) interval on repeated ECGs during RGT-419B monotherapy.

OTHER OUTCOMES:
Symptom Burden | through study completion, an average of 1 year
  Change from baseline in symptom burden on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) from baseline to end of treatment

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California, San Diego, La Jolla, California
  - University California, Los Angeles, Los Angeles, California
  - Hem-Onc Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - New York Cancer and Blood Specialists, Port Jefferson Station, New York